CLINICAL TRIAL: NCT00608179
Title: Glimepiride Induced Insulin Secretion Will be Inhibited by Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Steve Davis, Department Chair, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: IRB #020690
Record Dates: First submitted 2008-01-25; First posted 2008-02-06 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
Keywords: epinephrine; glucose clamp
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Glyburide; Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Glimepiride
- 2 (Experimental)
  Interventions: Drug: glyburide
- 3 (Experimental): control-euglycemia
  Interventions: Other: glucose clamp
- 4 (Experimental): control-hypoglycemia
  Interventions: Other: glucose clamp

INTERVENTIONS:
Drug: Glimepiride — Glimepiride (Amaryl) 4 mg oral dose during protocol, given once during each protocol.
  Other Names: Amaryl
  Arms: 1
Drug: glyburide — Glyburide (Dia-Beta) 10 mg oral dose during protocol, given once during each protocol.
  Other Names: Dia-Beta
  Arms: 2
Other: glucose clamp — Hyperinsulinemic euglycemic glucose clamp procedure-120 minutes
  Arms: 3
Other: glucose clamp — hypoglycemic glucose clamp procedure -120 minutes
  Arms: 4

SUMMARY:
This study will look at two FDA approved medications that improve how the pancreas works in patients with Type 2 Diabetes. In order to understand how these medications work in patients with diabetes we must first measure the normal response in healthy volunteers without diabetes. We will be looking at the body's normal physiological response to low blood sugar and whether this will be modified by these medicationsThe hypothesis would be that glimepiride induced insulin secretion will be inhibited by hypoglycemia.

DETAILED DESCRIPTION:
In patients with type 2 diabetes, sulfonylurea drugs are a mainstay for effective glucose control. These agents produce their hypoglycemic effects via stimulation of endogenous insulin secretion. Oversecretion of insulin, per se, or a continued relative increase of the hormone even when plasma glucose is normal will result in hypoglycemia. This latter situation commonly occurs if a patient decides to omit, delay, or reduce the size of a meal. An important defense against hypoglycemia in the above situations is glucose dependent regulation of insulin secretion. In other words, a low ambient glucose concentration could regulate the magnitude of the amount of insulin released in response to a sulfonylurea. Thus during hypoglycemic conditions, the sulfonylurea would result in little or no insulin secretion, whereas its effects during hyperglycemia would be amplified. Glimepiride and glyburide are both second-generation sulfonlyurea drugs used commonly for treatment of type 2 diabetes. This study will compare the two and ask the following question:

Is Glimepiride insulin secretion dependent upon glucose concentration in-vivo?

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 30-60
* Body Mass Index 21-30 kg/m2
* All potential volunteers will have routine blood test to screen for hepatic, renal, and hematological abnormalities
* EKG treadmill stress test for volunteers over 40 years of age.
* Female volunteers of childbearing potential will undergo HCG pregnancy test.

Exclusion Criteria:

* Prior or current history of poor health
* Abnormal results following screening tests
* Pregnancy
* History of allergy to sulfonylurea or related drugs

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2002-08; Primary Completion 2004-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
catecholamines | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University